CLINICAL TRIAL: NCT03820531
Title: DNA-mutation Analysis by Next Generation Sequencing in Cyst Fluid of Suspected Intraductal Papillary Mucinous Neoplasia of the Pancreas Obtained by Endoscopic Ultrasound-guided Fine Needle Aspiration (ZYSTEUS-Study)
Brief Title: DNA-mutation Analysis in Cyst Fluid of Suspected Intraductal Papillary Mucinous Neoplasia of the Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZYSTEUS-Study
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pancreas Cyst
Keywords: DNA Mutational Analysis; Cyst Fluid; Pancreas
MeSH Terms: conditions — Pancreatic Cyst | interventions — Cytological Techniques

STUDY DESIGN:
Intervention Model Description: DNA-mutation analysis by Next Generation Sequencing is performed to identify IPMN pancreas cysts with LGD versus HGD/Carcinoma.
  Controls: non-neoplastic pancreas cysts and chronic pancreatitis with main duct dilation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected mucinous pancreas cyst (Experimental): In all pancreas cysts > 15mm and/or pancreas duct dilatation > 5mm in patients who are fit for surgery EUS-guided pancreas cyst fluid aspiration is conducted. In cyst fluid CEA and lipase examination, cytology and Next Generation Sequencing is performed. After that, the pancreas cyst will be resected and histopathologically analysed.
  Interventions: Diagnostic Test: Next Generation Sequencing; Diagnostic Test: CEA and lipase; Diagnostic Test: Cytology; Diagnostic Test: Histology of resected pancreas cyst

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing — DNA Mutational Analysis in pancreas cyst fluid concerning KRAS/GNAS-mutations and mutations in tumor supressor genes
Diagnostic Test: CEA and lipase — Measuring CEA and lipase level in pancreas cyst fluid:
  CEA > 192 ng/ml and lipase > 200 U/l = mucinous cyst
Diagnostic Test: Cytology — Cytology in pancreas cyst fluid:
  mucinous versus non-mucinous cyst; LGD versus HGD/Carcinoma
Diagnostic Test: Histology of resected pancreas cyst — Histology of resected pancreas cyst concerning mucinous versus non-mucinous cyst, IPMN versus non-IPMN and LGD versus HGD/Carcinoma

SUMMARY:
Diagnostic tools are needed to identify mucinous cysts for further evaluation or follow-up respectively to identify cysts with HGD or invasive cancer at an early stage for surgical resection. Molecular genetic analysis of pancreatic cyst fluid is a new but rapidly evolving method to identify KRAS/GNAS oncogenic driver mutations in mucinous cysts and to identify tumour suppressor gene mutations which are involved in advanced cysts with HGD or carcinoma. The ongoing ZYSTEUS-study tries to implement DNA mutation analysis by Next Generation Sequencing in the diagnostic algorithm of pancreas cyst evaluation. The first aim is to distinguish mucinous from non-mucinous cysts. The second aim is to define relevant tumour suppressor gene mutations which are relevant to distinguish between LGD and HGD/carcinoma in mucinous cysts.

DETAILED DESCRIPTION:
Intraductal papillary mucinous neoplasm (IPMN) with low grade dysplasia (LGD) can progress to high grade dysplasia (HGD) or invasive cancer. Main duct IPMN, mixed type IPMN or branch duct IPMN with high risk stigmata are highly predictive for malignancy. Therefore, patients in good general state should be considered for surgical resection. Guidelines like the International Fukuoka Consensus Guidelines from 2017 or the European evidence-based Guidelines on Pancreatic cyst neoplasms from 2018 provide detailed recommendations on the management of IPMNs by focusing on clinical characteristics, image morphology, cytology and laboratory parameters. However, these applied guidelines still lead to surgical overtreatment of pancreas cysts based on the pathologic outcomes as neither HGD nor carcinoma is found in up to 82.1 % of the resected cysts. Cyst fluid sent for cytology usually provides adequate cellular material for analysis in only 31% of the cases and Endoscopic Ultrasound-guided forceps biopsy has not yet shown to be better than fine needle aspiration. Hence, further diagnostic tools are needed to identify mucinous cysts for further evaluation or follow-up respectively to identify cysts with HGD or invasive cancer at an early stage for surgical resection. Molecular genetic analysis of pancreatic cyst fluid is possibly able to identify KRAS/GNAS oncogenic driver mutations in mucinous cysts and to identify tumour suppressor gene mutations which are involved in advanced cysts with HGD or carcinoma. This workgroup described a high sensitive method of targeted Next Generation Sequencing in pancreas cyst fluid with a limit of detection of allele frequency down to 0.01 %. Further investigations of the ongoing ZYSTEUS-study are focused on the implementation of DNA mutation analysis by NGS in the diagnostic algorithm of pancreas cyst evaluation. The first aim is to reliably distinguish mucinous from non-mucinous cysts respectively main duct IPMN from chronic pancreatitis with main duct dilatation as the absence of KRAS/GNAS-mutations is highly predictive for non-mucinous diseases. The second aim is to define relevant tumour suppressor gene mutations which are relevant to differentiate LGD from HGD/carcinoma in mucinous cysts. DNA mutation analysis will be compared with already established peroperative diagnostic tests of pancreas cyst fluid: Measurement of CEA and lipase as well as cytology.

ELIGIBILITY:
Inclusion Criteria:

* pancreas cysts with cyst size > 15mm
* pancreas with main duct dilation > 5mm

Exclusion Criteria:

* patients who are not fit for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Patients with a mucinous pancreas cyst | From EUS-guided fine needle aspiration of pancreas cyst fluid up to seven days
  Number of patients with the preoperative diagnosis of a mucinous pancreas cyst (numerator) in correlation with the number of patients with a mucinous pancreas cyst confirmed by surgery (denominator)
Pancreas cyst with HGD or carcinoma | From EUS-guided fine needle aspiration of pancreas cyst fluid up to seven days
  Number of patients with the preoperative diagnosis of a HGD/carcinoma pancreas cyst (numerator) in correlation with the number of patients with a HGD/carcinoma pancreas cyst confirmed by surgery (denominator)

CONTACTS AND LOCATIONS:
Overall Officials: Christel Weiß, Prof.Dr., Study Chair — University of Heidelberg, Department of Medical Statistis
Locations (1):
- Tertiary referral hospital: Theresienkrankenhaus und St. Hedwig Hospital, Academic, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Felsenstein M, Noe M, Masica DL, Hosoda W, Chianchiano P, Fischer CG, Lionheart G, Brosens LAA, Pea A, Yu J, Gemenetzis G, Groot VP, Makary MA, He J, Weiss MJ, Cameron JL, Wolfgang CL, Hruban RH, Roberts NJ, Karchin R, Goggins MG, Wood LD. IPMNs with co-occurring invasive cancers: neighbours but not always relatives. Gut. 2018 Sep;67(9):1652-1662. doi: 10.1136/gutjnl-2017-315062. Epub 2018 Mar 2. PMID 29500184
- [Background] Kanda M, Sadakari Y, Borges M, Topazian M, Farrell J, Syngal S, Lee J, Kamel I, Lennon AM, Knight S, Fujiwara S, Hruban RH, Canto MI, Goggins M. Mutant TP53 in duodenal samples of pancreatic juice from patients with pancreatic cancer or high-grade dysplasia. Clin Gastroenterol Hepatol. 2013 Jun;11(6):719-30.e5. doi: 10.1016/j.cgh.2012.11.016. Epub 2012 Nov 28. PMID 23200980
- [Background] Singhi AD, McGrath K, Brand RE, Khalid A, Zeh HJ, Chennat JS, Fasanella KE, Papachristou GI, Slivka A, Bartlett DL, Dasyam AK, Hogg M, Lee KK, Marsh JW, Monaco SE, Ohori NP, Pingpank JF, Tsung A, Zureikat AH, Wald AI, Nikiforova MN. Preoperative next-generation sequencing of pancreatic cyst fluid is highly accurate in cyst classification and detection of advanced neoplasia. Gut. 2018 Dec;67(12):2131-2141. doi: 10.1136/gutjnl-2016-313586. Epub 2017 Sep 28. PMID 28970292
- [Background] Rosenbaum MW, Jones M, Dudley JC, Le LP, Iafrate AJ, Pitman MB. Next-generation sequencing adds value to the preoperative diagnosis of pancreatic cysts. Cancer Cytopathol. 2017 Jan;125(1):41-47. doi: 10.1002/cncy.21775. Epub 2016 Sep 20. PMID 27647802
- [Background] Amato E, Molin MD, Mafficini A, Yu J, Malleo G, Rusev B, Fassan M, Antonello D, Sadakari Y, Castelli P, Zamboni G, Maitra A, Salvia R, Hruban RH, Bassi C, Capelli P, Lawlor RT, Goggins M, Scarpa A. Targeted next-generation sequencing of cancer genes dissects the molecular profiles of intraductal papillary neoplasms of the pancreas. J Pathol. 2014 Jul;233(3):217-27. doi: 10.1002/path.4344. PMID 24604757
- [Background] Volckmar AL, Endris V, Gaida MM, Leichsenring J, Stogbauer F, Allgauer M, von Winterfeld M, Penzel R, Kirchner M, Brandt R, Neumann O, Sultmann H, Schirmacher P, Rudi J, Schmitz D, Stenzinger A. Next generation sequencing of the cellular and liquid fraction of pancreatic cyst fluid supports discrimination of IPMN from pseudocysts and reveals cases with multiple mutated driver clones: First findings from the prospective ZYSTEUS biomarker study. Genes Chromosomes Cancer. 2019 Jan;58(1):3-11. doi: 10.1002/gcc.22682. Epub 2018 Oct 17. PMID 30230086